CLINICAL TRIAL: NCT04999280
Title: Effect of Daily Consumption of a Fiber-enriched Croissant on Metabolic Status, Dietary Habits and Gut Microbiota in Healthy Subjects (CROMA)
Brief Title: Fiber-enriched Croissant Consumption and Effects on Metabolic Status, Appetite and Gut Microbiota
Acronym: CROMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Paola Vitaglione, Associate Professor, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CROMA
Record Dates: First submitted 2021-08-05; First posted 2021-08-10 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Healthy; Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fiber Croissant (FIBCRO) Group (Experimental): Daily consumption at breakfast for 2 weeks of a fiber-enriched croissant
  Interventions: Other: Fiber Croissant (FIBCRO) Group
- Control Croissant (CONCRO) Group (Active Comparator): Daily consumption at breakfast for 2 weeks of a control croissant
  Interventions: Other: Control Croissant (CONCRO) Group

INTERVENTIONS:
Other: Fiber Croissant (FIBCRO) Group — Subjects will consume for 2 weeks at breakfast a fiber-enriched sourdough croissant. All subjects will be requested not to change other dietary habits and their physical activity during the 2 week intervention period.
  Other Names: Fiber-enriched Croissant
  Arms: Fiber Croissant (FIBCRO) Group
Other: Control Croissant (CONCRO) Group — Subjects will consume for 2 weeks at breakfast a sourdough croissant. All subjects will be requested not to change other dietary habits and their physical activity during the 2 week intervention period.
  Other Names: Control Croissant
  Arms: Control Croissant (CONCRO) Group

SUMMARY:
The aim of this study is to evaluate the effect of a daily consumption for 2 weeks of a sourdough croissant enriched with dietary fibers vs a control sourdough croissant with no fiber added on daily energy intakes, fasting metabolic parameters, inflammatory status, blood pressure, anthropometric measures, body composition, appetite sensations, gastrointestinal functionality and gut microbiota composition.

DETAILED DESCRIPTION:
Associations between human health, diet and gut microbiota composition and functionality have been widely highlighted by the scientific literature in this field. Evidence shows that population adopting a Western dietary model, with a reduced intake of dietary fiber, undergo an adaptation of the gut microbiota characterized by the loss of some bacterial species and a general reduction in microbial biodiversity. The national guidelines for a healthy diet suggest to include daily fruit, vegetables, whole grains and legumes (the main sources of fiber in the diet) in the habitual diet to reduce the risk of diseases and to improve health. However, the compliance with these nutritional recommendations is generally low among individuals. Therefore, the commercial availability of dietary fiber-enriched products could be advantageous.

Breakfast is an important meal that should provide at least 20% of the daily calories with an adequate supply of all nutrients. Having fiber-enriched foods for breakfast could bring numerous nutritional benefits and if they are made with sourdough may be even better. Indeed, sourdough leavened baked products provide compounds with potential prebiotic activity, reduce the glucose and insulin response, increase satiety and reduce gastro-intestinal disorders upon consumption.

The hypothesis is that the combination of sourdough and dietary fiber in baked products could further ameliorate glucose metabolism in consumers compared to sourdough products.

The aim of this study is to evaluate the effects of a daily consumption at breakfast for 2 weeks of a sourdough croissant enriched with dietary fibers from 10 different sources vs a sourdough croissant with no fiber added (control) on daily energy intakes, metabolic and inflammatory status, appetite feelings, body weight, body mass index (BMI), waist and hip circumferences, body composition, blood pressure, gut microbiota composition and gastrointestinal functionality in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects;
* men and women;
* age 18-50 years;
* 20 kg/m2 ≤ BMI ≤ 35 kg/m2;
* habitual daily breakfast consumption (≥ 250kcal/day);
* habitual diet characterized by absence of any food supplements and alternative medication, probiotics and prebiotics, whole grain and/or fiber enriched foods;
* intake of fruit/vegetables < 3 servings/day;
* low level of physical activity;
* signed written informed consent.

Exclusion Criteria:

* food allergies and intolerances and celiac disease;
* gastrointestinal diseases;
* relevant diseases;
* pregnant or breastfeeding;
* previous abdominal surgery;
* hypertriglyceridemia (Triglycerides > 200 mg/dL);
* hypercholesterolemia (Total cholesterol > 200 mg/dL);
* hyperglycaemia (glycaemia ≥ 110 mg/dL);
* hypertension (arterial blood pressure ≥140/90 mm Hg);
* weight loss ≥ 3 kg within 2 months before the study;
* antibiotics treatment within 3 months before the study;
* any medication (different from antibiotics) at the enrollment and within 2 months before the study;
* habitual diet characterized by high fruit and vegetables intakes (>3 portion/die);
* high level of physical activity;
* alcohol consumption ≥ 3 alcohol units per day;
* simultaneous participation in other trial.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Variation of daily energy intakes | 2 weeks
  Calculation of total daily energy intakes based on 7 days food records

SECONDARY OUTCOMES:
Changes in fasting plasma inflammatory markers | 2 weeks
  Measure of plasma C-reactive protein (mmol/L)
Changes in fasting plasma lipids | 2 weeks
  Measure of plasma concentrations (mg/dL) of Total-, LDL-, and HDL-Cholesterol, as well as Triglycerides
Changes in fasting blood glucose | 2 weeks
  Measure of blood glucose concentrations (mg/dL)
Variation of serum Insulin hormone concentration | 2 weeks
  Measure of serum Insulin concentrations (mg/dL)
Variation of plasma endocannabinoids and N-acyl-ethanolamines concentration | 2 weeks
  Measure of plasma endocannabinoids and N-acyl-ethanolamines concentrations (mg/dL)
Variation of serum dipeptidyl-dipeptidase-IV activity | 2 weeks
  Measure of serum dipeptidyl-dipeptidase-IV (U/L) activity
Variation of urinary excretion levels of polyphenols | 2 weeks
  Measure of polyphenols concentration in urine by mean of liquid chromatography coupled with tandem mass spectrometry (LC/MS/MS)
Variation of urinary excretion levels of urolithins | 2 weeks
  Measure of urolithins concentration in urine by mean of LC/MS/MS
Changes in stool consistency | 2 weeks
  Measure of consistency of feces by mean of King's stool chart filled out by subjects. The chart comprises four categories of stool consistency: hard and formed, soft and formed, loose and unformed, liquid.
Changes in stool weight | 2 weeks
  Measure of stool weight by mean of King's stool chart filled out by subjects. The chart comprises three categories of stool weight : <100 g, 100-200 g, >200 g.
Changes in stool frequency | 2 weeks
  Measure of frequency of feces by mean of King's stool chart filled out by subjects. Fecal frequency is incorporated by recording the code of each feces passed over a 24 hour period.
Changes in gastrointestinal functionality | 2 weeks
  Calculation of daily fecal score from summation of all scores for stool consistency, weight and frequency obtained from King's stool chart filled out by subjects. Scores are weighted such that an increase in fecal frequency alone results in a higher score than a change in fecal consistency alone, which in turn results in a higher score than an increase in fecal weight alone. Diarrhea is classified by a daily fecal score of 15 or more.
Changes in faecal microbiome | 2 weeks
  The composition of faecal microbiome will be determined by high throughput sequencing of the ribosomal ribonucleic acid 16S (16S rRNA) gene. The massive number of sequences obtained will be analyzed by using state of the art bioinformatics tools and the presence and relative abundance of the microbial species occurring in each sample will be determined.
Changes in body weight | 2 weeks
  Measure of body weight in fasting subjects
Changes in body mass index | 2 weeks
  Calculation of body mass index by using the formula weight in kilograms divided by height in meters squared.
Changes in waist circumference | 2 weeks
  Measure of waist circumference at the midpoint between the lower margin of the least palpable rib and the top of the iliac crest.
Changes in hip circumference | 2 weeks
  Measure of hip circumference around the widest portion of the buttocks.
Changes in blood pressure | 2 weeks
  Measure of systolic pressure and diastolic pressure in millimetres of mercury (mmHg) by using a digital sphygmomanometer
Changes in body composition | 2 weeks
  Body composition is determined by conventional bioelectrical impedance analysis with a single-frequency 50 kilohertz (kHz) bioelectrical impedance analyzer in the postabsorptive state (fasting subjects) and after being in the supine position for 20 min. Body composition data will be calculated from bioelectrical measurements and anthropometric data by using validated predictive equations.
Variation of hunger feeling scores | 2 weeks
  Measures of hunger sensation over the day reported by subjects by using hunger Visual Analogue Scales (VAS) 0-10 centimeters (where 0 corresponds to the lowest and 10 to the highest feeling the individual could perceive). Changes in these scores may reflect potential effects of dietary intervention in modulating hunger.
Variation of fullness feeling scores | 2 weeks
  Measure of fullness sensation over the day reported by subjects by using fullness Visual Analogue Scales (VAS) 0-10 centimeters (where 0 corresponds to the lowest and 10 to the highest feeling the individual could perceive). Changes in these scores may reflect potential effects of dietary intervention in modulating fullness.
Variation of satiety feeling scores | 2 weeks
  Measure of satiety sensation over the day reported by subjects by using satiety Visual Analogue Scales (VAS) 0-10 centimeters (where 0 corresponds to the lowest and 10 to the highest feeling the individual could perceive). Changes in these scores may reflect potential effects of dietary intervention in modulating satiety.

CONTACTS AND LOCATIONS:
Overall Officials: Paola Vitaglione, Professor, Study Director — Department of Agricultural Sciences, Federico II University
Locations (1):
- Department of Agricultural Sciences, Federico II University, Portici, Italy

REFERENCES:
- [Derived] Barone Lumaga R, Tagliamonte S, De Rosa T, Valentino V, Ercolini D, Vitaglione P. Consumption of a Sourdough-Leavened Croissant Enriched with a Blend of Fibers Influences Fasting Blood Glucose in a Randomized Controlled Trial in Healthy Subjects. J Nutr. 2024 Oct;154(10):2976-2987. doi: 10.1016/j.tjnut.2024.08.015. Epub 2024 Aug 22. PMID 39179206